CLINICAL TRIAL: NCT03556579
Title: The Effects of Contact Lenses With Experimental Dye on Visual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6100
Record Dates: First submitted 2018-05-31; First posted 2018-06-14 (Actual); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): For Visit 1, subjects will be randomly assigned to 1 of 2 contralateral lens sequences (Right: Test, Left: Control) OR (Right: Control, Left: Test). Then for visit 2, subjects will be randomly assigned to the same 1 of 2 contralateral lens sequences again.
  Interventions: Device: senofilcon A with new UV blocker; Device: senofilcon A
- Control/Test (Experimental): For Visit 1, subjects will be randomly assigned to 1 of 2 contralateral lens sequences (Right: Test, Left: Control) OR (Right: Control, Left: Test). Then for visit 2, subjects will be randomly assigned to the same 1 of 2 contralateral lens sequences again.
  Interventions: Device: senofilcon A with new UV blocker; Device: senofilcon A

INTERVENTIONS:
Device: senofilcon A with new UV blocker — Test Lens
Device: senofilcon A — Control Lens

SUMMARY:
This is a single-site, two-visit, contralateral, non-dispensing, randomized, controlled and subject-masked study to measure potential benefits of the new UV blocker.

ELIGIBILITY:
Inclusion Criteria:

- Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol
3. Between 18 and 65 (inclusive) years of age at the time of screening.
4. Be a current spherical soft silicone hydrogel contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week wear time over the last 30 days by self-report.
5. The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 through -4.50 D in each eye.
6. The subject has a best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or breastfeeding.
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any autoimmune disease or use of medication, which may interfere with contact lens wear. Habitual medications used by successful soft contact lens wearers are considered acceptable.
4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.
5. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Multifocal, toric or extended wear contact lens correction.
8. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
9. History of binocular vision abnormality or strabismus.
10. Any infectious disease (e.g., hepatitis, tuberculosis) or contagious immunosuppressive diseases (e.g., HIV) by self-report.
11. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
12. Any ocular infection.
13. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia Center for Sight, Statesboro, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 62 subjects were into this study. Of those enrolled, 60 were assigned and administered a study lens. Two subjects were enrolled but not administered a study lens. All 60 subjects completed the study.
Pre-assignment Details: Subjects were stratified into two age groups: 18-39 and 40-65 using a 2:1 allocation. Subjects were randomized at each visit using a contralateral design.
Groups:
- OD:Test, OS:Control/ OD:Test, OS:Control: Subjects that were randomized to receive the Test lens in their right eye and the Control lens in their left eye at both visit 1 and visit 2.
- OD:Test, OS:Control/ OD:Control, OS:Test: Subjects that were randomized to receive at visit 1 the Test lens in their right eye and the Control lens in their left eye and at visit 2 was randomized to receive the Control lens in their right eye and the Test lens in their left eye.
- OD:Control, OS:Test/ OD:Test, OS:Control: Subjects that were randomized to receive at visit 1 the Control lens in their right eye and the Test lens in their left eye and at visit 2 was randomized to receive the Test lens in their right eye and the Control lens in their left eye.
- OD:Control, OS:Test/ OD:Control, OS:Test: Subjects that were randomized to receive the Control lens in their right eye and the Test lens in their left eye at both visit 1 and visit 2.
Period: Visit 1
Arm/Group | OD:Test, OS:Control/ OD:Test, OS:Control | OD:Test, OS:Control/ OD:Control, OS:Test | OD:Control, OS:Test/ OD:Test, OS:Control | OD:Control, OS:Test/ OD:Control, OS:Test
Started | 16 | 14 | 14 | 16
Completed | 16 | 14 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Visit 2
Arm/Group | OD:Test, OS:Control/ OD:Test, OS:Control | OD:Test, OS:Control/ OD:Control, OS:Test | OD:Control, OS:Test/ OD:Test, OS:Control | OD:Control, OS:Test/ OD:Control, OS:Test
Started | 16 | 14 | 14 | 16
Completed | 16 | 14 | 14 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: All Subjects that were Fit with at least one study lens.
Arm/Group | Safety Population
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 11
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  American Indian or Alaska Native | 1
  Black or African American | 22
  White | 35
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Two-Point Light Spread Function
Description: The two-point light spread function was assessed at visit 2 for each subject eye under two conditions with a distance filter and without a distance filter. Measurements for this metric were taken twice, with the presence of an additional UV/HEV light source and without this additional light source (the same study lenses were used for both measurements). Two-point light spread function is defined that the as the minimum distance (mm) that two points of light are completely distinct. Measurements for this metric are positive. Smaller distances indicate better lens performance. The average distance for each lens type and light source combination was reported across age groups.
Time Frame: Between 5 minutes and 3 hours Post Lens Insertion, at Visit 2
Population: All subjects that completed the study without a major protocol deviation impacting any primary endpoint.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Groups:
- Testing With Additional Light Source: Subjects that wore the Test lens in either eye during visit 2. This lens was measured using an additional light source.
- Control With Additional Source: Subjects that wore the Control lens in either eye during visit 2. This lens was measured using an additional light source.
- Test Without Additional Light Source: Subjects that wore the Test lens in either eye during visit 2. This lens was measured without using an additional light source.
- Control Without Additional Light Source: Subjects that wore the Control lens in either eye during visit 2. This lens was measured without using an additional light source.
Arm/Group | Testing With Additional Light Source | Control With Additional Source | Test Without Additional Light Source | Control Without Additional Light Source
Number analyzed (Participants) | 54 | 54 | 54 | 54
Number analyzed (Eyes) | 54 | 54 | 54 | 54
mm
  with distance filter | 5.36 (3.132) | 6.71 (2.521) | 6.47 (3.304) | 7.48 (3.149)
  Without Dustance Filter | 2.29 (1.129) | 3.37 (1.214) | 3.05 (1.205) | 3.78 (1.472)
Statistical Analysis 1: Comparison: Test Without Additional Light Source vs Control Without Additional Light Source; Without Distance Filter; Test type: Superiority — Superiority was concluded if the upper limit of the 95% confidence interval was below 0. No sample size calculation was performed for this study since historical data was not available for either study lens for any of the primary endpoints; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.01 to -0.36], Standard Error of Mean 0.162 — Mean difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Testing With Additional Light Source vs Control With Additional Source; Without Distance Filter; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-1.45 to -0.81], Standard Error of Mean 0.162 — Mean difference was calculated as Test - Control

2. Primary Outcome: Halos
Description: The appearance of Halos was assessed at visit 2 for each subject eye. Measurements for this metric were taken twice, with the presence of an additional UV/HEV light source and without this additional light source (the same study lenses were used for both measurements). Halos were quantified as the diameter (mm) of the outer edges of the Halo. Measurements for this metric are positive. Smaller diameter indicates better lens performance. The average diameter (mm) for each lens type and light source combination was reported across age groups.
Time Frame: Between 5 minutes and 3 hours Post Lens Insertion, at Visit 2
Population: All subjects that completed the study without a major protocol deviation impacting any primary endpoint.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Testing With Additional Light Source | Control With Additional Source | Test Without Additional Light Source | Control Without Additional Light Source
Number analyzed (Participants) | 54 | 54 | 54 | 54
Number analyzed (Eyes) | 54 | 54 | 54 | 54
mm | 29.20 (15.777) | 52.57 (22.758) | 39.09 (14.524) | 46.73 (18.355)
Statistical Analysis 1: Comparison: Test Without Additional Light Source vs Control Without Additional Light Source; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = -8.86, 95% CI 2-sided [-13.16 to -4.55], Standard Error of Mean 2.173 — Mean difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Testing With Additional Light Source vs Control With Additional Source; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = -24.93, 95% CI 2-sided [-29.24 to -20.62], Standard Error of Mean 2.173 — Mean difference was calculated as Test - Control

3. Secondary Outcome: Glare Disability Threshold
Description: The Glare disability threshold was assessed for each eye at visit 1. The study lenses in this visit were assessed without the additional light sourced used at visit 2. Subjects were exposed to a target stimulus for 2 seconds; before the measurement was taken the annulus was set to a level below that which would cause the target stimulus to be veiled. The experimenter would then adjust the intensity of the annulus until subjects could no longer see the target stimulus. Subjects would indicate this by pressing a buzzer. Glare disability thresholds take on positive values, where higher values indicate better lens performance. The average glare disability level (change in log relative energy) for each lens type was reported across age groups.
Time Frame: Between 5 minutes and 3 hours Post Lens Insertion, at Visit 1
Population: All subjects that completed the study without a major protocol deviation impacting any primary endpoint.
Measure: Mean (Standard Deviation); unit: log units
Units Other Than Participants: eyes
Arm/Group | Test Without Additional Light Source | Control Without Additional Light Source
Number analyzed (Participants) | 54 | 54
Number analyzed (eyes) | 54 | 54
log units | 0.98 (0.166) | 1.16 (0.140)
Statistical Analysis 1: Comparison: Test Without Additional Light Source vs Control Without Additional Light Source; Test type: Superiority — Superiority was concluded if the lower limit of the 95% confidence interval was above 0. No sample size calculation was performed for this study since historical data was not available for either study lens for any of the primary endpoints; Linear Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.15 to 0.23], Standard Error of Mean 0.022 — Mean Difference was calculated as Test minus Control

4. Secondary Outcome: Photostress Recovery Time
Description: Photostress Recovery (PR) Time (seconds) was assessed for each eye at visit 1. The study lenses in this visit were assessed without the additional light sourced used at visit 2. Subjects are exposed to a target, once the target was able to be comfortable viewed by the subject, a bright bleaching light covered it. As the afterimage fades, participants will gradually be able to re-gain sight of the target. PR time will be recorded as the time it takes following exposure to the bleaching light to regain sight of the target. PR Times are positive values where smaller times indicate better lens performance. The average PR Time (seconds) for each lens type was reported across age groups.
Time Frame: Between 5 minutes and 3 hours Post Lens Insertion, at Visit 1
Population: Subjects that completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Test Without Additional Light Source | Control Without Additional Light Source
Number analyzed (Participants) | 54 | 54
Number analyzed (eyes) | 54 | 54
seconds | 8.83 (8.668) | 17.28 (15.230)
Statistical Analysis 1: Comparison: Test Without Additional Light Source vs Control Without Additional Light Source; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Generalized linear mixed model; Generalized Linear mixed model with a lognormal distribution using the Kenward and Roger method for the denominator degrees of freedom; Mean Ratio = 0.55, 95% CI 2-sided [0.46 to 0.65]

5. Secondary Outcome: Glare Discomfort
Description: The Glare discomfort (change in palpebral fissure height) was assessed for each eye at visit 1. The study lenses in this visit were assessed without the additional light sourced used at visit 2. Glare discomfort can take on negative and positive values, where smaller values indicate better lens performance. The average glare discomfort (change in palpebral fissure height) for each lens type was reported across age groups.
Time Frame: Between 5 minutes and 3 hours Post Lens Insertion, at Visit 1
Population: Subjects that completed all study visits wihtout a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Test Without Additional Light Source | Control Without Additional Light Source
Number analyzed (Participants) | 54 | 54
Number analyzed (eyes) | 54 | 54
mm | 2.26 (1.249) | 2.90 (1.569)
Statistical Analysis 1: Comparison: Test Without Additional Light Source vs Control Without Additional Light Source; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-1.07 to -0.15], Standard Error of Mean 0.230 — Mean Difference was calculated as Test minus Control

6. Secondary Outcome: Heterochromatic Contrast Threshold
Description: Heterochromatic Contrast Threshold was assessed for each eye at visit 1. The study lenses in this visit were assessed without the additional light sourced used at visit 2. Heterochromatic contrast thresholds are measured as thresholds to a variable wavelength central target presented on a short-wave (460nm) sky-light background. Thresholds are positive values, where higher values indicate better lens performance. The average threshold each lens type was reported across age groups.
Time Frame: Between 5 minutes and 3 hours Post Lens Insertion, at Visit 1
Population: Subjects that completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: log units
Units Other Than Participants: eyes
Arm/Group | Test Without Additional Light Source | Control Without Additional Light Source
Number analyzed (Participants) | 54 | 54
Number analyzed (eyes) | 54 | 54
log units | 1.01 (0.170) | 1.24 (0.164)
Statistical Analysis 1: Comparison: Test Without Additional Light Source vs Control Without Additional Light Source; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Linear Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.14 to 0.23], Standard Error of Mean 0.022 — Mean Difference was calculated as Test minus Control

7. Primary Outcome: Starburts
Description: The appearance of starbursts was assessed at visit 2 for each subject eye. Measurements for this metric were taken twice, with the presence of an additional UV/HEV light source and without this additional light source (the same study lenses were used for both measurements). Starbursts are defined as the diameter (mm) of the light's lateral spread. Measurements for this metric are positive. Smaller diameter indicates better lens performance. The average diameter (mm) for each lens type and light source combination was reported across age groups.
Time Frame: Between 5 minutes and 3 hours Post Lens Insertion, at Visit 2
Population: Subjects that have completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Testing With Additional Light Source | Control With Additional Source | Test Without Additional Light Source | Control Without Additional Light Source
Number analyzed (Participants) | 54 | 54 | 54 | 54
Number analyzed (eyes) | 54 | 54 | 54 | 54
mm | 45.66 (24.228) | 75.12 (27.370) | 55.78 (23.037) | 69.60 (25.914)
Statistical Analysis 1: Comparison: Testing With Additional Light Source vs Control With Additional Source; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = -30.56, 95% CI 2-sided [-31.66 to -25.46], Standard Error of Mean 2.555 — Mean difference was calculated as Test minus Control
Statistical Analysis 2: Comparison: Test Without Additional Light Source vs Control Without Additional Light Source; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = -15.38, 95% CI 2-sided [-20.48 to -10.27], Standard Error of Mean 2.555 — Mean difference was calculated as Test Minus Control

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. One to 14 days per subject.
Groups:
- Test: All subjects that wore the Test lens at either visit 1 or visit 2.
- Control: All subjects that wore the Control lens at either visit 1 or visit 2.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT03556579/Prot_SAP_000.pdf